CLINICAL TRIAL: NCT04520269
Title: A Single Arm, Phase Ib/II Trial of Single Agent Pacritinib in Patients With 1q21.3 Amplified Solid Tumors Enriching for Interleukin-1 Receptor-associated Kinase 1 (IRAK1) Pathway Activation (PAIR)
Brief Title: A Single Arm, Phase Ib/II Trial of Single Agent Pacritinib in Patients With 1q21.3 Amplified Solid Tumors Enriching for Interleukin-1 Receptor-associated Kinase 1 Pathway Activation (PAIR)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC02/04/19
Record Dates: First submitted 2020-08-11; First posted 2020-08-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: 1q21.3; interleukin-1 receptor-associated kinase 1; Pacritinib; IRAK1
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, lead in phase Ib dose confirmation, followed by phase II study with 2 parallel study cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with (cfDNA) 1q21.3 copy number amplification (Experimental): The phase Ib segment will be carried out in a standard 3+3 design. In the phase II portion, 2 parallel cohorts will be enrolled (Cohort A: 1q21.3 amplified breast cancers, Cohort B: 1q21.3 amplified other solid tumors).
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — 3+3 design Dose Level 1 :200mg BD every 4 weeks Dose Level -1 :200mg OM, 100mg ON every 4 weeks Dose Level -2 :100mg BD every 4 weeks

SUMMARY:
This is a single arm, open-label, lead in phase Ib dose confirmation, followed by phase II study with 2 parallel study cohorts. Patients will be pre-screened for presence of 1q21.3 copy number amplification in plasma samples prior to screening process. Only patients with confirmed plasma cell-free DNA (cfDNA) 1q21.3 copy number amplification who successfully meet study eligibility criteria will be enrolled.

The phase Ib segment will be carried out in a standard 3+3 design, with a projected enrolment of 3 to 18 patients to determine the RP2D. In the phase II portion, 2 parallel cohorts will be enrolled (Cohort A: 1q21.3 amplified breast cancers, Cohort B: 1q21.3 amplified other solid tumors). Based on the Simon 2 stage optimal design, 12 patients will be enrolled in each cohort for stage I of the study, and assessed for PFS. If at least 3 of 12 patients meet study response criteria, the study will then be expanded to stage 2 to include a total of 25 patients in each cohort. Accounting for 10% attrition rate, a maximum of 28 patients will be enrolled into each cohort for phase II of the study.

DETAILED DESCRIPTION:
2.1. Hypothesis

* Single agent pacritinib is effective in disease control of patients with 1q21.3 amplified solid tumors
* Single agent pacritinib is safe in patients with 1q21.3 amplified solid tumors
* Treatment with pacritinib will decrease plasma cfDNA copy number ratio of 1q21.3 in patients with 1q21.3 amplified solid tumors
* Plasma cfDNA copy number ratio of 1q21.3 will correlate with serial radiological findings in patients with 1q21.3 amplified solid tumors

2.2. Primary Objectives

• To determine the proportion of patients with 1q21.3 amplified breast cancer (primary population: Cohort A) who remain progression-free at 4 months after treatment with pacritinib

2.3. Secondary Objectives

* To determine the safety and tolerability of pacritinib in patients with treatment refractory solid tumors
* To determine the RP2D of pacritinib in patients with treatment refractory solid tumors
* To evaluate disease response from pacritinib by RECIST criteria version 1.1 and tumor markers
* To determine the proportion of patients with 1q21.3 amplified treatment refractory solid tumors excluding (exploratory population: Cohort B) who remain progression-free at 4 months after treatment with pacritinib

2.4. Exploratory Objectives

* To determine pharmacokinetic (PK) parameters including Cmax/min and steady state concentrations of pacritinib through serial plasma sampling
* To determine pharmacodynamics (PD) parameters including highly sensitive C-reactive protein (CRP), HbA1c, changes in cytokine levels and plasma cfDNA levels of copy number ratio of 1q21.3
* Correlation of plasma cfDNA levels of copy number ratio of 1q21.3 with radiological findings determined by RECIST criteria 1.1 and tumor markers

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

* Age > or = 21 years.
* Histological or cytological diagnosis of malignant advanced solid tumors refractory to standard therapy or for which no suitable effective standard therapy exists.

  o Patients who fit above criteria will be pre-screened for presence of 1q21.3 amplification using a plasma assay based on digital PCR. Patients with tumors that exhibit 1q21.3amplification will be enrolled. Positive 1q21.3 amplification is defined as more than 3 standard deviations above the mean comparing the averaged copy number ratio of 3 genes (TUFT1, S100A8 and S100A7) relative to the reference gene RPP30 measure in sample (13).
* ECOG 0-2
* Has measureable or evaluable disease based on RECIST 1.1 criteria
* Estimated life expectancy of at least 12 weeks.
* Has documented progressive disease from last line of therapy
* Has recovered from acute toxicities from prior anti-cancer therapies
* Adequate organ function including the following:

  * Bone marrow:

    * Absolute neutrophil (segmented and bands) count (ANC) > or = 1.5 x 109/L
    * Platelets > or = 100 x 109/L
    * Hemoglobin > or = 8 x 109/L
  * Hepatic:

    * Bilirubin < or = 1.5 x upper limit of normal (ULN),
    * ALT or AST < or = 2.5x ULN, (or < or = 5 X with liver metastases)
  * Renal:

    * Creatinine < or = 1.5x ULN
* Signed informed consent from patient
* Able to comply with study-related procedures.
* Prior therapy (patients enrolled in phase Ib may be enrolled if they fulfil prior therapy criteria for either Cohort A or Cohort B)

  * Cohort A only: Has received at least 2 lines of systemic therapy (endocrine or chemotherapy) in the palliative setting. Chemotherapy in an adjuvant setting for which patients relapsed within 6 months of completion can be considered as line(s) of palliative therapy.
  * Cohort B only: Any number of prior lines of palliative chemotherapy.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Significant recent bleeding history defined as CTCAE grade 2 or higher within the past 3 months, unless precipitated by an inciting event (e.g. surgery, trauma, injury).
* Suboptimal cardiac function, defined by:

  * Any history of CTCAE grade > or = 2 non-dysrhythmia cardiac conditions within the last 6 months
  * New York Heart Association class II, III or IV congestive cardiac failure
  * Left ventricular ejection fraction of <45%
* QTc prolongation of >450ms as assessed by ECG or other factors that increase the risk of QT interval prolongation
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Unable to comply with study procedures
* Systemic treatment with a strong CYP3A4 inhibitor or storn CYP450 inducer within 14 days prior to treatment Day 1

Phase Ib lead-in can recruit patients who fulfil critieria for either Cohort A or Cohort B AND all other inclusion/exclusion criteria

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall radiological response rate | 36 months
  Rates of radiological response (complete and partial clinical response), including confidence intervals. measured by RECIST 1.1
Progression-free survival | 36 months
  Proportion of patients in cohort A and Cohort B who remain progression-free at 4 months
Overall safety of pacritinib in patients with treatment refractory solid tumors | 36 months
  Safety measures that will be used in the study include physical examinations and clinical laboratory tests (haematology and blood chemistries). Patients will be rated for toxicity during each cycle of treatment using the NCI CTCAE scale, version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Joline Si Jing Lim, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caswell-Jin JL, Plevritis SK, Tian L, Cadham CJ, Xu C, Stout NK, Sledge GW, Mandelblatt JS, Kurian AW. Change in Survival in Metastatic Breast Cancer with Treatment Advances: Meta-Analysis and Systematic Review. JNCI Cancer Spectr. 2018 Nov;2(4):pky062. doi: 10.1093/jncics/pky062. Epub 2018 Dec 24. PMID 30627694
- [Background] Crown J, Dieras V, Kaufmann M, von Minckwitz G, Kaye S, Leonard R, Marty M, Misset JL, Osterwalder B, Piccart M. Chemotherapy for metastatic breast cancer-report of a European expert panel. Lancet Oncol. 2002 Dec;3(12):719-27. doi: 10.1016/s1470-2045(02)00927-0. PMID 12473512